CLINICAL TRIAL: NCT01611688
Title: First Human Dose Trial of NNC0215-0384 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8210-3926; 2011-003008-19 (EudraCT Number); U1111-1122-3474 (Other: WHO)
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid | interventions — NNC0215-0384

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: NNC0215-0384
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0215-0384 — I.v.(intravenous) dose-escalation. Highest dose planned for i.v. administration is 10 mg/kg
  Arms: Active
Drug: placebo — Administered i.v.(intravenous) or s.c. (subcutaneous, under the skin).
  Arms: Placebo
Drug: NNC0215-0384 — The s.c. (subcutaneous, under the skin) part will not start until at least two i.v. dose levels have been evaluated for safety and pharmacokinetics. Highest dose planned for s.c. administration is 4 mg/kg
  Arms: Active

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to describe the safety and tolerability of single intravenous (i.v.) and subcutaneous (s.c.) doses of NNC0215-0384 in subjects with active rheumatoid arthritis (RA) on background methotrexate (MTX) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Active RA, characterised by a DAS28 (CRP)(Disease Activity Score based on 28 joints and CRP) above 3.2 and a minimum of two swollen joints based on a 68/66 joint count at screening
* Concomitant treatment with MTX (7.5 - 25 mg/week both inclusive) for at least 16 weeks, with a stable dose for at least 6 weeks prior to dosing

Exclusion Criteria:

* Subjects with chronic inflammatory autoimmune disease other than RA
* History of or current inflammatory joint disease other than RA such as gout (crystal proven), psoriatic arthritis, juvenile idiopathic arthritis, current reactive arthritis or Lyme disease
* Any active or ongoing chronic infectious disease (e.g. chronic osteomyelitis, chronic pyelonephritis) requiring systemic anti-infectious treatment within 4 weeks prior to randomisation
* Clinically significant cardiac or cardiovascular disease
* Past or current malignancy
* Latent or active tuberculosis (TB) as documented by: A positive QuantiFeron® test (test can be performed up to 2 months prior to dosing). One retest is allowed in case of inconclusive results.- A history of active TB within the last 3 years even, if treated effectively. - A history of active TB more than 3 years ago, if there is no documentation that the prior anti-TB treatment was appropriate in duration and type

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06-04 (Actual); Primary Completion 2013-06-17 (Actual); Study Completion 2013-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 10 weeks after trial product administration

SECONDARY OUTCOMES:
I.v. administration: AUC, Area under the curve | Up to 10 weeks after drug administration
I.v. administration: terminal half-life (t½) | Up to 10 weeks after drug administration
S.c. administration: AUC, Area under the curve | Up to 10 weeks after drug administration
S.c. administration: terminal half-life (t½) | Up to 10 weeks after drug administration
Maximum level and duration of full C5a receptor (C5aR) occupancy by NNC0215-0384 on neutrophils | Up to 10 weeks after drug administration
Maximum and minimum levels of relevant serum and plasma biomarkers related to NNC0215-0384 safety, efficacy or mechanism of action (MoA) | Up to 10 weeks after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com